CLINICAL TRIAL: NCT00684177
Title: A Randomized, Double-Blind, Multicenter, Placebo-controlled, Phase III Superiority Study to Assess the Safety and Efficacy of Topical Retapamulin Ointment, 1%, Versus Placebo Ointment Applied Twice Daily for 5 Days in the Treatment of Adult and Pediatric Subjects With SITL
Brief Title: Retapamulin Versus Placebo in Secondarily-Infected Traumatic Lesions (SITL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOC110977
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Skin Infections, Bacterial
Keywords: infection; retapamulin; secondarily-infected traumatic lesions; placebo
MeSH Terms: conditions — Cellulitis; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retapamulin Ointment, 1% (Experimental)
  Interventions: Drug: Retapamulin Ointment, 1%
- Placebo Ointment (Placebo Comparator)
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: Retapamulin Ointment, 1% — Provided as approximately 10 grams of an off-white smooth ointment in collapsible aluminum tubes with reverse taper puncture tip caps.
  Other Names: Retapamulin Ointment; 1%
  Arms: Retapamulin Ointment, 1%
Drug: Placebo ointment — Provided as approximately 10 grams of an off-white smooth ointment in collapsible aluminum tubes with reverse taper puncture tip caps.
  Arms: Placebo Ointment

SUMMARY:
The purpose of Study TOC110977 is to demonstrate clinical superiority of Retapamulin ointment, 1%, over placebo in patients with secondarily-infected traumatic lesions, which includes secondarily-infected lacerations, abrasions and sutured wounds. Subjects 2 months of age and older will be treated with topical retapamulin or placebo ointment twice daily for 5 days. The primary endpoint of this study is the clinical response at follow-up (Day 12-14; 7-9 days after the end of therapy) in the intent-to-treat clinical population.

DETAILED DESCRIPTION:
This is a prospective, multicenter, double-blind, placebo-controlled parallel group study in subjects aged 2 months and older with SITL, including secondarily-infected lacerations, sutured wounds or abrasions. A laceration or sutured wound cannot exceed 10 cm in length with surrounding erythema not extending more than 2 cm from the edge of the lesion. Abrasions cannot exceed 100 cm2 in total area, or up to a maximum of 2% total body surface area for subjects <18 years of age, with surrounding erythema not extending more than 2 cm from the edge of the abrasion.

There are four study visits occurring over a 12-14 day period. At the Baseline visit (Visit 1, Day 1), subjects will be randomized to receive retapamulin or placebo ointment in a 2:1 (retapamulin:placebo) ratio. The 2:1 randomization is included to minimize the number of subjects exposed to treatment with placebo. Both active treatment and placebo will be dosed topically twice daily (BID) for 5 days. All subjects will receive a telephone call from the investigator or appropriate designee appointed by the investigator on Day 2. The subject will be interviewed to determine if there is any evidence of worsening infection. Subjects who are thought to be worsening will be instructed to come in to the clinic for an assessment. Subjects will be monitored and clinically evaluated at the On-therapy (Days 3-4), End of Therapy (Days 7-9), and Follow-up (Days 12-14) visits.

Randomization will be center-based and performed using an appropriate Interactive Voice Response System (IVRS), an automated telephone system. The block size will remain confidential.

Subjects are considered to have completed the study if they meet all inclusion/exclusion criteria, are considered compliant with study medication, and attend all study visits as defined by the protocol.

ELIGIBILITY:
Inclusion criteria:

* subject is aged 2 months or older
* subject has secondarily-infected traumatic lesion (laceration, sutured wound or abrasion)
* negative urine pregnancy test
* subject has total skin infection rating scale score of at least 8, including pus/exudate score of at least 3
* subject and/or parent/legal guardian is willing and able to comply with protocol
* subject or parent/legal guardian has given written informed consent or assent as applicable

Exclusion criteria:

* previous hypersensitivity to pleuromutilin
* secondarily-infected animal/human bite or puncture wound
* subject has an abscess
* chronic ulcerative lesion
* underlying skin disease
* systemic signs and symptoms of infection
* infection not appropriately treated with topical antibiotic
* infection requires surgical intervention prior to or during study
* subject received systemic antibacterial or steroid, or topical therapeutic agent within 24 hours of entry into study
* serious underlying disease
* subject pregnant, breast feeding or planning a pregnancy, or unacceptable method of contraception
* other investigational drug within 30 days of study entry
* subject previously enrolled in this study

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (51):
- United States (30):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Arlington Heights, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Teaneck, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Norristown, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Vienna, Virginia
- Argentina (4):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Chivilocoy, Buenos Aires
  - GSK Investigational Site, Loma Hermosa, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Brazil (3):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Curitiba/Paraná, Paraná
  - GSK Investigational Site, Passo Fundo, Rio Grande do Sul
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vadodara
  - GSK Investigational Site, Wardha
- South Africa (9):
  - GSK Investigational Site, Belville
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Hatfield
  - GSK Investigational Site, Lynnwood
  - GSK Investigational Site, Midrand
  - GSK Investigational Site, Newton
  - GSK Investigational Site, Welkom
  - GSK Investigational Site, Worcester

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TOC110977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 508 participants were randomized. One participant did not receive treatment; thus, no data were collected for this participant. Only 507 participants were included in the analysis.
Groups:
- Retapamulin: Topical retapamulin ointment, 1% twice daily for 5 days
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Retapamulin | Placebo
Started | 343 | 164
Completed | 322 | 141
Not Completed | 21 | 23
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 10 | 15
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retapamulin | Placebo | Total
Number analyzed (Participants) | 343 | 164 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (18.77) | 28.6 (18.32) | 31.3 (18.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 63 | 207
  Male | 199 | 101 | 300
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 144 | 71 | 215
  American Indian or Alaskan Native | 9 | 3 | 12
  Asian - Central / South Asian Heritage | 0 | 1 | 1
  Asian - East Asian Heritage | 4 | 2 | 6
  Asian - South East Asian Heritage | 33 | 15 | 48
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 132 | 61 | 193
  Mixed Race | 19 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success and Failure at Follow-up (7-9 Days Post Therapy) for the Primary Efficacy Population
Description: "Clinical Success" at follow-up was defined as "Resolution of clinically meaningful signs and symptoms of infection recorded at baseline including a pus/exudate Skin Infection Rating Scale (SIRS) score of "0". Clinical response at follow-up was classified as "Clinical Failure" for all other cases. The SIRS consists of seven items (pus/exudates, crusting, erythema/inflammation, tissue warmth, tissue edema, itching and pain). Each item has a score ranging from 0 to 6 (0=absent, 6=severe). The SIRS total score was calculated as the sum of the scores of all 7 SIRS items.
Time Frame: Days 12-14
Population: Primary Efficacy Population: ITTC participants (par.) with baseline pus/exudate >=3 who were enrolled under the original protocol with data captured under eCRF V1 and who were enrolled under protocol amendments with data captured under eCRF V2; ITTC (Intent-to-treat Clinical): all randomized par. who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 246 | 113
participants
  Clinical Success | 184 | 75
  Clinical Failure | 62 | 38
Statistical Analysis 1: Comparison: Retapamulin vs Placebo; Test type: Superiority or Other; p = 0.098, Chi-squared; Risk Difference (RD) = 8.4, 95% CI 2-sided [-1.6 to 18.4]

2. Secondary Outcome: Number of Participants With Clinical Success and Failure at Follow-up (7-9 Days Post Therapy) for the Intent-to-Treat Bacteriology (ITTB) Subset of the Primary Efficacy Population
Description: as for outcome 1
Time Frame: Days 12-14
Population: ITTB subset of Primary Efficacy Population: participants in the Primary Efficacy Population (see analysis population description in the Primary Outcome section) who had at least one pathogen isolated at the baseline visit.
Measure: Number; unit: participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 182 | 84
participants
  Clinical Success | 139 | 54
  Clinical Failure | 43 | 30
Statistical Analysis 1: Comparison: Retapamulin vs Placebo; Test type: Superiority or Other; p = 0.04, Chi-squared; Risk Difference (RD) = 12.1, 95% CI 2-sided [0.6 to 23.6]

3. Secondary Outcome: Number of Participants With Microbiological Success and Failure at Follow-up (7-9 Days Post Therapy)
Description: The "by pathogen" microbiological outcome was determined by comparing the baseline culture results to those at follow-up. The "by subject" microbiological response was "Microbiological Success" if the microbiological outcomes for all baseline pathogens (bps) belong to "Eradication" (elimination of bps), "Presumed Eradication" (clinical outcome was success; no culture was obtained due to lack of culturable material), or "Colonization" (previously unidentified pathogen is identified at end of therapy in participant who is resolved/improved); otherwise, response was "Microbiological Failure".
Time Frame: Days 12-14
Population: ITTB subset of Primary Efficacy Population
Measure: Number; unit: participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 182 | 84
participants
  Microbiological Success | 139 | 54
  Microbiological Failure | 43 | 30
Statistical Analysis 1: Comparison: Retapamulin vs Placebo; Test type: Superiority or Other; p = 0.04, Chi-squared; Risk Difference (RD) = 12.1, 95% CI 2-sided [0.6 to 23.6]

4. Secondary Outcome: Number of Participants With the Indicated Clinical Outcome at End of Therapy (2-4 Days Post Therapy)
Description: Clinical outcome is determined by the investigator based on signs and symptoms (S/S) at the end of therapy evaluation. The 4 clincal outcome categories are: clinical success, resolution of clinically meaningful S/S of infection recorded at baseline (BL), including a pus/exudates score of 0; clinical improvement, improvement of S/S of infection recorded at BL to such an extent that no further antimicrobial therapy is necessary; clinical failure, insufficient improvement of deterioration of S/S of infection recorded at BL such that additional antibiotic therapy is required; unable to determine.
Time Frame: Days 7-9
Population: Primary Efficacy Population
Measure: Number; unit: participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 246 | 113
participants
  Clinical Success | 130 | 52
  Clinical Improvement | 102 | 45
  Clinical Failure | 11 | 14
  Unable to Determine | 3 | 2

5. Secondary Outcome: Number of Baseline Pathogens With the Indicated Microbiological Outcome at End of Therapy (2-4 Days Post Therapy)
Description: The "by pathogen" microbiological outcome was determined by comparing the baseline culture results to those at follow-up. The results presented below pooled all baseline pathogens (bps). Eradication: elimination of bps. Presumed Eradication: clinical outcome was success; no culture was obtained due to lack of culturable material. Presumed Improvement: clinical outcome was improvement such that no culture was obtained due to lack of culturable material. Persistence: bps still present. Presumed persistence: clinical failure and no culture was obtained.
Time Frame: Days 7-9
Population: ITTB subset of Primary Efficacy Population
Measure: Number; unit: baseline pathogens
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 243 | 110
baseline pathogens
  Eradication | 4 | 5
  Presumed Eradication | 137 | 49
  Presumed Improvement | 94 | 35
  Persistence | 3 | 13
  Presumed Persistence | 5 | 8

6. Secondary Outcome: Number of Participants With Therapeutic Success and Failure at Follow-up (7-9 Days Post Therapy)
Description: "Therapeutic Success (Succ)" was referred to as both "Clinical Succ" and "Microbiological (Micro) Succ" at Follow-up. "Clinical Succ" was the "Resolution of baseline signs/symptoms of infection with a pus score of "0." A participant was "Micro Succ" if the micro outcome for all baseline pathogens (bps) belonged to "Eradication" (elimination of bps), "Presumed Eradication" (clinical outcome is success; no culturable material), or "Colonization" (new pathogen is identified at end of therapy in participants who are resolved/improved). All other combinations were deemed "Therapeutic Failures."
Time Frame: Follow-up (Days 12-14)
Population: ITTB subset of Primary Efficacy Population
Measure: Number; unit: participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 182 | 84
participants
  Success | 139 | 54
  Failure | 43 | 30

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the first dose of study medication until study completion. Serious AEs (SAEs) were collected from the time of consent and continued until study completion (including the Follow-up Period).
Description: AEs were collected for all randomized participants (par.) who received at least one dose of study medications (i.e., ITTC Population). Safety data were analyzed based on the actual treatment received. One par. who was randomized to retapamulin treatment but actually received placebo was included in the placebo arm for the safety analyses.
Arm/Group | Retapamulin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/342 | 1/165
Other Adverse Events (participants affected / at risk) | 8/342 | 4/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin (N=342) | Placebo (N=165)
Myocardial infarction (Cardiac disorders) | 1 | 0
Pneumococcal pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin (N=342) | Placebo (N=165)
Application site pain (General disorders) | 5 | 0
Condition aggravated (General disorders) | 3 | 1
Pyrexia (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.